CLINICAL TRIAL: NCT02004236
Title: Transcranial Random Noise Noninvasive Brain Stimulation Applied to the Fronto-temporal Cortex Improves Verbal Fluency and Emphaty in Children With Autistic Spectrum Disorder
Brief Title: Fronto-temporal tDCS Mproves Fluency & Empathy in ASD Kids
Acronym: tDCS25112013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Foundation for Neurometrics Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Autism and tDCS
Record Dates: First submitted 2013-11-25; First posted 2013-12-09 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Autism; ASD
Keywords: tDCS; QEEG; ERP; ASD; Autism; verbal fluency; empathy; noninvasive brain stimulation
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tRNS Fronto-temporal cortex (Experimental): This group receive 35 sessions of tRNS over fronto-temporal cortex
  Interventions: Device: tRNS Fronto-temporal cortex
- tRNS over fusiform temporal cortex (Experimental): This group receive 35 sessions of tRNS over fusiform temporal cortex
  Interventions: Device: tRNS over fusiform temporal cortex
- tRNS with sham (Placebo Comparator): This group receive 35 sessions with sham
  Interventions: Device: tRNS with sham

INTERVENTIONS:
Device: tRNS Fronto-temporal cortex — This group receive 35 sessions of tRNS over fronto-temporal cortex
  Arms: tRNS Fronto-temporal cortex
Device: tRNS over fusiform temporal cortex — This group receive 35 sessions of tRNS over fusiform temporal cortex
  Arms: tRNS over fusiform temporal cortex
Device: tRNS with sham — the subjects receive 35 session with sham
  Arms: tRNS with sham

SUMMARY:
Interventional, prospective, randomized, double-blind, placebo-controlled and parallel assignment study, in which patients with Autism Spectrum Disorder (ASD) are two types of intervention by transcranial random noise stimulation (tRNS), to improve verbal fluency and empathy.

DETAILED DESCRIPTION:
Interventional, prospective, randomized, double-blind, placebo-controlled and parallel assignment study, in which patients receive three types of intervention tRNS: one group received 35 sessions focused on the fronto-temporal cortex, another group received 35 sessions focused on the temporal fusiform cortex and last placebo group was operated with 35 sessions tRNS. After brain noninvasive stimulation sessions, a blind analysis of the improvement in verbal fluency and empathy in patients with autism spectrum disorder is made. For each patient included a follow up period of three months will be established.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 5 and 12 years.
* Meet DSM-IV criteria for autism spectrum disorder.
* Patients who have been diagnosed at least 2 years before inclusion in the study.

Exclusion Criteria:

* Acute visual or hearing loss.
* Traumatic brain injury.
* Other neurological disorders: migraine, epilepsy, tuberous sclerosis ...
* Trauma at birth.
* Mental retardation.
* Pregnancy.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Neville, MD, Principal Investigator — New Remedies Ltd
Locations (2):
- United Kingdom (2):
  - New Remedies Ltd, Liverpool, Merseyside
  - Moises Aguilar Domingo, Liverpool, Spain

REFERENCES:
- See also: Bigdata4brain LTD — https://www.bigdata4brain.co.uk/

RESULTS

PARTICIPANT FLOW:
Groups:
- tRNS Over Fronto-temporal Cortex: This group receive 35 sessions of tRNS over fronto-temporal cortex
  tRNS Fronto-temporal cortex: This group receive 35 sessions of tRNS over fronto-temporal cortex
Period: Overall Study
Arm/Group | tRNS Over Fronto-temporal Cortex | tRNS Over Fusiform Temporal Cortex | tRNS With Sham
Started | 75 | 75 | 75
Completed | 75 | 75 | 59 (Leave the group because the parents does't find any clinical improvement.)
Not Completed | 0 | 0 | 16
Not completed — Lack of Efficacy | 0 | 0 | 16

BASELINE CHARACTERISTICS:
Population: Clinically referred sample of young children between 5 and 12 years old with ASD
Groups:
- Total: Total of all reporting groups
Arm/Group | tRNS Fronto-temporal Cortex | tRNS Over Fusiform Temporal Cortex | tRNS With Sham | Total
Number analyzed (Participants) | 75 | 75 | 59 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (1.98) | 6.9 (2.1) | 7.2 (2.3) | 7.2 (2.12)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 75 | 75 | 59 | 209
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Customized [Mean (Standard Deviation); unit: years]
  4-6 years | 5.1 (0.80) | 4.8 (1.17) | 5.3 (0.75) | 5.06 (0.91)
  7-9 years | 7.2 (0.9) | 8.4 (0.73) | 7.8 (1.1) | 7.8 (0.91)
  10-12 years | 11.2 (0.48) | 10.1 (0.69) | 10.8 (0.88) | 10.7 (0.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 75 | 75 | 59 | 209
Region of Enrollment [Number; unit: participants]
  Spain | 75 | 75 | 59 | 209

OUTCOME MEASURES:

1. Primary Outcome: Verbal Fluency
Description: Goal: Improve in verbal fluency in ASD children between 5 and 12 years. We use D-KEFS (Delis-Kaplan Executive Function System Delis Kaplan Sorting Test), Verbal Fluency Subtest - Category Condition.
  Description: The verbal fluency Category test evaluates fluent productivity in the verbal domain by asking participants to generate exemplars belonging to the category animals, and subsequently, boys´ names. Participants were given 60 s to do it.
  Values: Category scores were based on the average number of items generated in the two categories (animals and boys´names) during 60 s.
  Time Frame: Baseline (Before treatment) and 1 day Post-treatment (after completing 3 months of intensive speech therapy during tRNS sessions)
Time Frame: During 3 months of intensive speech therapy during tRNS sessions
Population: Time frame: Baseline Before treatment and after completing 3 months of intensive speech therapy during tRNS sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tRNS Fronto-temporal Cortex | tRNS Over Fusiform Temporal Cortex | tRNS With Sham
Number analyzed (Participants) | 75 | 75 | 59
units on a scale
  before tRNS | 9.3 (1.3) | 10.5 (1.6) | 9.9 (1.1)
  after tRNS | 8.3 (1.2) | 10.4 (1.1) | 10 (0.9)

2. Primary Outcome: Sociability
Description: Goal: Evaluate emphaty with CARS scale in autism spectrum disorder children between 5 and 12 years after tRNS sessions.
  CARS (Childhood Autism Rating Scale) by Shopler & Reichler (1971) in Spanish version EVAI (Escala de Valoración de Autismo Infantil) by Leal-Soto, F.; Aguirre, L.P. y Williams, E.E.
  Description: 15 items in the scale that evaluate: Relating to people, Imitative Behavior, Emotional Response, Body Use, Object Use, Adaptation to Change, Visual Response, Listening Response, Perceptive Response, Fear or Anxiety, Verbal Communication, Non-Verbal Communication, Activity level, Level and consistency of Intellective Relations and General Impressions.
  Values: The CARS scores range from 15 to 60, with lower scores indicating better outcome. It classifies the child as not autistic (below 30), moderately autistic (30-36.5) or severely autistic (above 36.5)
Time Frame: During 3 months of intensive speech therapy during tRNS sessions
Population: Time frame: Baseline Before treatment and after completing 3 months of intensive speech therapy during tRNS sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tRNS Fronto-temporal Cortex | tRNS Over Fusiform Temporal Cortex | tRNS With Sham
Number analyzed (Participants) | 75 | 75 | 59
units on a scale
  before tRNS | 30.6 (1.9) | 32.1 (2.2) | 31.8 (3.4)
  after tRNS | 19.4 (2.1) | 20.2 (1.8) | 30.1 (2.5)

3. Secondary Outcome: Ratio Theta/Beta Before tDCS
Description: The purpose of the present study was to determine if the theta/beta ratio, and theta and beta separately, correlate with behavioral parameters, and if these measures discriminate between children a with Autism Spectrum disorder (ASD) and normal gender- and age-matched controls before and after tRNS intervention in ASD children between 5 and 12 years old.
Time Frame: During 3 months of intensive speech therapy during tRNS sessions
Measure: Mean (Standard Deviation); unit: Ratio theta/beta before tRNS
Groups:
- tDCS Fronto-temporal Cortex: This group receive 35 sessions of tRNS over fronto-temporal cortex
  tRNS Fronto-temporal cortex: This group receive 35 sessions of tRNS over fronto-temporal cortex
- tDCS Over Fusiform Temporal Cortex: This group receive 35 sessions of tRNS over fusiform temporal cortex
  tRNS over fusiform temporal cortex: This group receive 35 sessions of tRNS over fusiform temporal cortex
- tDCS With Sham: This group receive 35 sessions with sham
  tRNS with sham: the subjects receive 35 session with sham
Arm/Group | tDCS Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
Ratio theta/beta before tRNS | 25 (0.88) | 30 (1.1) | 26 (0.53)

4. Secondary Outcome: Theta Amplitude in T5 Before tDCS
Description: as for outcome 3
Time Frame: During 3 months of intensive speech therapy during tRNS sessions
Measure: Mean (Standard Deviation); unit: MicroVolts
Groups:
- tDCS Over Fronto-temporal Cortex: This group receive 35 sessions of tRNS over fronto-temporal cortex
  tRNS Fronto-temporal cortex: This group receive 35 sessions of tRNS over fronto-temporal cortex
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
MicroVolts | 3.2 (0.3) | 2.7 (0.11) | 3.5 (0.5)

5. Secondary Outcome: Ratio Theta/Beta After tDCS
Description: The purpose of the present study was to determine if the theta/beta ratio, and theta and beta separately, correlate with behavioral parameters, and if these measures discriminate between children a with Autism Spectrum disorder (ASD) and normal gender- and age-matched controls before and after tDCS intervention in ASD children between 5 and 12 years old.
Time Frame: During 3 months of intensive speech therapy during tDCS sessions
Measure: Mean (Standard Deviation); unit: Ratio theta/beta after tRNS
Groups:
- tDCS Over Fronto-temporal Cortex: This group receive 35 sessions of tDCS over fronto-temporal cortex
  ttDCS Fronto-temporal cortex: This group receive 35 sessions of tDCS over fronto-temporal cortex
- tDCS Over Fusiform Temporal Cortex: This group receive 35 sessions of tDCS over fusiform temporal cortex
  tDCS over fusiform temporal cortex: This group receive 35 sessions of tDCS over fusiform temporal cortex
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tRNS With Sham
Number analyzed (Participants) | 75 | 75 | 59
Ratio theta/beta after tRNS | 12 (1.1) | 14 (0.52) | 25 (0.77)

6. Secondary Outcome: Theta Amplitude in T5 After tDCS
Description: Evaluate QEEG (brainwave changes in frequency bandfs and amplitude) after tRNS intervention in ASD children between 5 and 12 years old
Time Frame: During 3 months of intensive speech therapy during tRNS sessions
Measure: Mean (Standard Deviation); unit: MicroVolts
Groups:
- tDCS Over Fronto-temporal Cortex: This group receive 35 sessions of tDCS over fronto-temporal cortex
  tDCS Fronto-temporal cortex: This group receive 35 sessions of tDCS over fronto-temporal cortex
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
MicroVolts | 2.2 (0.41) | 1.5 (0.36) | 3.3 (0.84)

7. Secondary Outcome: Reaction Time in ECPT Before tDCS
Description: ERP & Behaviour changes in ASD children after tDCS
Time Frame: During 3 months of intensive speech therapy during tRNS sessions
Measure: Mean (Standard Deviation); unit: Milliseconds
Groups:
- tDCS With Sham: This group receive 35 sessions with sham
  tDCS with sham: the subjects receive 35 session with sham
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
Milliseconds | 756 (23.5) | 698 (34.2) | 722 (18.9)

8. Secondary Outcome: Omission Errors Before tDCS
Description: ERP and behaviour changes in ASD children before tDCS
Time Frame: During 3 months of intensive speech therapy during tRNS sessions
Measure: Mean (Standard Deviation); unit: number of errors during ECPT task
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
number of errors during ECPT task | 85 (5.2) | 91 (3.2) | 88 (4.6)

9. Secondary Outcome: Commission Errors Before tDCS
Description: ERP and Behaviour changes in ASD children before tDCS
Time Frame: During 3 months of intensive speech therapy during tDCS sessions
Measure: Median (Standard Deviation); unit: number of omission errors VCPT task
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
number of omission errors VCPT task | 6 (0.2) | 8 (1.1) | 19 (0.9)

10. Secondary Outcome: P3b Wave Amplitude Before tDCS
Description: ERP and behaviour Changes in ASD children before tDCS
Time Frame: During 3 months of intensive speech therapy during tRNS sessions
Measure: Mean (Standard Deviation); unit: MicroVolts or Amplitude P3b wave
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
MicroVolts or Amplitude P3b wave | 0.5 (0.12) | 0.7 (0.4) | 0.3 (0.2)

11. Secondary Outcome: Reaction Time After tDCS
Description: ERP and behaviour Changes in ASD children after tDCS
Time Frame: During 3 months of intensive speech therapy during tDCS sessions
Measure: Mean (Standard Deviation); unit: Reaction Time measuring in Milliseconds
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
Reaction Time measuring in Milliseconds | 690 (10.4) | 556 (7.4) | 714 (3.2)

12. Secondary Outcome: Omissions Errors After tDCS
Description: ERP and behaviour Changes in ASD children after tDCS
Time Frame: During 3 months of intensive speech therapy during tDCS sessions
Measure: Mean (Standard Deviation); unit: number of omission errors in VCPT task
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 75
number of omission errors in VCPT task | 68 (2.3) | 57 (4.7) | 20 (1.8)

13. Secondary Outcome: Commission Errors After tDCS
Description: ERP and behaviour Changes in ASD children after tDCS
Time Frame: During 3 months of intensive speech therapy during tDCS sessions
Measure: Mean (Standard Deviation); unit: number of commission errors in VCPT task
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
number of commission errors in VCPT task | 6 (0.2) | 8 (1.1) | 19 (0.9)

14. Secondary Outcome: P3b Wave Amplitude After tDCS
Description: ERP and behaviour Changes in ASD children after tDCS
Time Frame: During 3 months of intensive speech therapy during tDCS sessions
Measure: Mean (Standard Deviation); unit: MicroVolts or Amplitude P3b wave
Arm/Group | tDCS Over Fronto-temporal Cortex | tDCS Over Fusiform Temporal Cortex | tDCS With Sham
Number analyzed (Participants) | 75 | 75 | 59
MicroVolts or Amplitude P3b wave | 2.1 (0.25) | 1.8 (0.65) | 0.4 (0.32)

ADVERSE EVENTS:
Arm/Group | tRNS Fronto-temporal Cortex | tRNS Over Fusiform Temporal Cortex | tRNS With Sham
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75 | 0/59
Other Adverse Events (participants affected / at risk) | 1/75 | 2/75 | 0/59
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tRNS Fronto-temporal Cortex (N=75) | tRNS Over Fusiform Temporal Cortex (N=75) | tRNS With Sham (N=59)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) — The children are disorientated in time and space at least during 1 or 2 hours after tRNS session

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less